CLINICAL TRIAL: NCT05881291
Title: Efficacy and Safety of Ciprofol for General Anaesthesia in Patients Undergoing Transcatheter Aortic Valve Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0135
Record Dates: First submitted 2023-05-15; First posted 2023-05-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2024-07

CONDITIONS: Hemodynamics; Transcatheter Aortic Valve Replacement; General Anesthesia; Post-induction Hypotension
Keywords: ciprofol; transcatheter aortic valve replacement; general anesthesia
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Alfentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group ciprofol (Experimental): Patients receive ciprofol for general anesthesia
  Interventions: Drug: ciprofol
- group propofol (Active Comparator): Patients receive propofol for general anesthesia
  Interventions: Drug: propofol

INTERVENTIONS:
Drug: ciprofol — induction of anesthesia：group ciprofol received an IV injection of ciprofol at a dose of 0.2-0.4 mg/kg, and administration time of 30 s.When the eyelash reflex disappeared and the BIS value was ≤60 administration was stopped, followed by an IV injection of alfentanil 30 μg/kg and rocuronium 0.6 mg/kg.
  Maintenance of anesthesia: group ciprofol received an IV infusion of ciprofol 0.8-2.4 mg·kg-1·h-1.
  Other Names: alfentanil
  Arms: group ciprofol
Drug: propofol — induction of anesthesia：group propofol received an IV injection of propofol at a dose of 1.0-2.0 mg/kg, and administration time of 30 s. When the eyelash reflex disappeared and the BIS value was ≤60 administration was stopped, followed by an IV injection of alfentanil 30 μg/kg and rocuronium 0.6 mg/kg.
  Maintenance of anesthesia:group propofol received an IV infusion of propofol 4-6 mg·kg-1·h-1.
  Other Names: alfentanil
  Arms: group propofol

SUMMARY:
Aortic valve stenosis is the most common debilitating valvular heart lesion in old patients. Transcatheter aortic valve replacement (TAVR) is an emergent technique for high-risk patients with aortic stenosis. In recent times, treatment has expanded to also include low- and intermediate-risk individuals. General anesthesia offers many advantages, mainly regarding the possibility of an early diagnosis and treatment of possible complications through the use of transesophageal echocardiography. Propofol is the most used sedative-hypnotic agent for the induction and maintenance of general anesthesia. However, adverse events such as hypotension, and bradycardia are associated with propofol sedation. Ciprofol is a novel anesthetic/sedative agent similar to propofol, with an equivalent efficacy ratio to propofol of 1/4 to 1/5. Ciprofol has properties of fast onset of action, rapid recovery, reduced injection pain and stable cardiorespiratory function, making it a promising alternative to propofol. The aim of this study is to explore the safety and efficacy of ciprofol when used for general anesthesia in patients undergoing transcatheter aortic valve replacement compared to propofol.

DETAILED DESCRIPTION:
After assessing patient eligibility, they were randomly assigned to two equally sized groups.Patients in this study were fasted for a minimum of 8 h without premedication.

Following arrival in the operating room, patients were monitored with electrocardiography, respiratory rate, pulse oximetry, bispectral index (BIS), cerebral oxygen saturation,and continuous invasive arterial blood pressure. Induction of anesthesia： group ciprofol received an IV injection of ciprofol at a dose of 0.2-0.4 mg/kg, and administration time of 30 s； group propofol received an IV injection of propofol at a dose of 1.0-2.0 mg/kg, and administration time of 30 s.

When the eyelash reflex disappeared and the BIS value was ≤60 administration was stopped, followed by an IV injection of alfentanil 30 μg/kg and rocuronium 0.6 mg/kg.

Endotracheal intubation was performed when alfentanil and rocuronium had fully worked, and the BIS value was <50. A ventilator was then connected for mechanical ventilation using the following parameters: VT 6-8 ml/kg, RR 12-20 times/min, the inspiratory-to-expiratory ratio of 1:2, oxygen flowed 2 L/min, and maintaining PETCO2 at 35-45 mmHg (1 mmHg=0.133 kPa).

Maintenance of anesthesia:

group ciprofol received an IV infusion of ciprofol 0.8-2.4 mg·kg-1·h-1； group propofol received an IV infusion of propofol 4-6 mg·kg-1·h-1 .

ELIGIBILITY:
Inclusion Criteria:

* patients planned for transfemoral transcatheter aortic valve replacement
* expected duration of surgery ≥ 1 and ≤ 3h
* patients undergoing general anesthesia
* no gender limit，age≥60 years，≤85 years
* BMI ≥18 and ≤30kg/m2
* ASA physical status 3~4
* be able to understand the procedures and methods of the trial and voluntarily sign the informed consent form

Exclusion Criteria:

* predicted presence of difficult airway or previous history of difficult airway
* allergic to eggs, soy products, propofol, and opioids and their antidotes
* patients with shock or hypotension that is difficult to correct with vasopressor
* patients with mental, nervous system diseases, long-term use of sedatives or antidepressants
* HB < 10.0 g/dL (100 g/L)
* patients with previous long-term use of sedative and analgesic drugs
* patients with severe heart，lung，liver and kidney disease
* not suitable for participation in this study as assessed by the investigator

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
primary endpoint was the area under the curve below baseline MAP (MAP-time integral) during the 15 min after induction | from the start of induction of anesthesia to 15 minutes after induction of anesthesia
  the area under the baseline MAP over the first 15 min after induction, called the MAP-time integral

SECONDARY OUTCOMES:
Incidence of hypotension | within 15 minutes after induction of anesthesia
  Hemodynamic variable
Incidence of bradycardia | within 15 minutes after induction of anesthesia
  Hemodynamic variable
dose of vasopressor used within 15 minutes after induction of anesthesia and vasopressor drugs used during surgery | during the surgery
  Hemodynamic variable
Incidence of injection pain | during the induction of anesthesia procedure
  injection pain
Incidence of postoperative nausea and vomiting | 1 day (during anesthesia awakening)
  drug reaction
Quality of life and disease recovery (QoR-15) score on postoperative day 1 | 1 day after surgery
  postoperative evaluation
changes of IL-6 before and one first day after surgery | immediately before surgery and one first day after surgery
  inflammatory factor level
changes of CK-MB and cTnT before and one first day after surgery | immediately before surgery and one first day after surgery
  myocardial enzyme level
Composite Clinical Endpoint at 1 Year (Extended Follow-up Analysis) | 1 year post-procedure
  The composite endpoint is defined as the occurrence of all-cause mortality, stroke, acute kidney injury (AKI), myocardial infarction (MI), or new-onset atrial fibrillation (NOAF). This is a post-hoc extended analysis. While the original trial protocol focused on intraoperative hemodynamics, these long-term data were prospectively collected via the institutional TAVR registry. The analysis of these 1-year outcomes was authorized under a specific ethical approval (No. 2025-1849) obtained after the primary trial completion.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Ni T, Zhou X, Wu S, Lv T, Hu Y, Gao Q, Luo G, Xie C, Zou J, Chen Y, Zhao L, Xiao J, Tao X, Yi Y, Xu Z, Wang T, Zhou J, Yao Y, Yan M. Hemodynamic Impact of Cipepofol vs Propofol During Anesthesia Induction in Patients With Severe Aortic Stenosis: A Randomized Clinical Trial. JAMA Surg. 2025 Jul 1;160(7):763-770. doi: 10.1001/jamasurg.2025.1299. PMID 40397427